CLINICAL TRIAL: NCT07027345
Title: A Phase II, Closed Label, Placebo Controlled, Randomized, Double-Blinded Clinical Trial to Evaluate the Efficacy and Safety of TolaSure Gel, 5% w/w Targeting Aggregated Mutant Keratin in Epidermolysis Bullosa Simplex (TAMES)
Brief Title: A Phase II, Placebo Controlled, Clinical Trial of Topical TolaSure Targeting Aggregated Mutant Keratin in Epidermolysis Bullosa Simplex
Acronym: (TAMES)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioMendics, LLC (Industry)
Collaborators: Northwestern University Feinberg School of Medicine (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Stanford University (Other); Lucile Packard Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAMES-02
Record Dates: First submitted 2025-06-09; First posted 2025-06-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Epidermolysis Bullosa Simplex
Keywords: Epidermolysis Bullosa; Epidermolysis Bullosa Simplex; EBS; Severe EBS; EBS Dowling-Meara; EBS Koebner; Skin Diseases; Keratin; Aggregate; Mutant; EBS-DM; Keratin Disorder; Skin Abnormalities; generalized; intermediate
MeSH Terms: conditions — Epidermolysis Bullosa Simplex; Epidermolysis Bullosa; Skin Diseases; Skin Abnormalities

STUDY DESIGN:
Intervention Model Description: Part 1 of the study (2-months total) will involve a randomized, double-blinded treatment assignment model where one arm will receive active, and the other arm will receive placebo. Part 2 of the study (2-months total) will involve a single arm crossover where the placebo arm will crossover and receive active. The active arm will continue treating with active. During this part of the study the treatment labels will still be blinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5% TolaSure Topical Gel (Active Comparator): 5% (w/w) TolaSure Gel
  Interventions: Drug: 5% TolaSure Topical Gel
- Topical Placebo Gel (Placebo Comparator): Placebo Control Gel
  Interventions: Drug: Topical Placebo Gel

INTERVENTIONS:
Drug: 5% TolaSure Topical Gel — TolaSure Topical Gel is applied once-daily to designated treatment areas for up to 4 months (Part 2 End of Study).
  Arms: 5% TolaSure Topical Gel
Drug: Topical Placebo Gel — Topical Placebo Gel is applied once-daily to designated treatment areas for up to 2 months (Part 1 End of Study).
  Arms: Topical Placebo Gel

SUMMARY:
This Phase II clinical study will assess the efficacy, safety and tolerability of topical TolaSure Gel in adults and pediatric patients (4 years of age and older) diagnosed with generalized intermediate to severe epidermolysis bullosa simplex (EBS). Each patient (40 to complete) will be enrolled in the study and will be randomized to receive either TolaSure Gel or a topical Placebo for daily application for 2-months. After 2-months, all patients will receive TolaSure Gel to daily apply for an additional 2-months. A remote follow-up visit will occur 2-months after the end of study. Total time in the study is 6-months. Patients will be applying study medication to randomized treatment area(s) (a minimum of ~2-3% Body Surface Area (BSA)), with the option to treat their feet as well throughout the study.

DETAILED DESCRIPTION:
This is a closed-label, Phase II clinical study to assess the efficacy, safety and tolerability of the investigational product (IP), topical TolaSure Gel, 5% w/w, in adults and pediatric patients diagnosed with generalized intermediate to severe epidermolysis bullosa simplex (EBS). TolaSure Gel, 5% w/w and Placebo tubes will be placed into kits where all labels (tubes and kit labels) will be blinded for drug content. Kits will be bundled (based on expected amount of study gel usage) and distributed randomly to patients [Goal of patient population, 1:1 M:F and approximately 70% pediatric patients].

Each patient (40 to complete) will be enrolled in the study and once a blistering flare is confirmed by the clinical study team, and the patient will be randomized to receive either TolaSure Gel, 5% w/w or Placebo (50:50 chance).

For Part 1 of the study, daily application of randomized treatment for 2 months will be applied to selected Target Lesional Areas (TLAs; a minimum area of approximately 2-3% Body Surface Area (BSA)). If a TLA resolves completely the patient will continue to treat designated area(s). Additionally, patients have the option to daily treat their feet.

For Part 2 of the study, a single arm crossover will then allow those patients that received Placebo to go on TolaSure Gel, 5% w/w for a subsequent 2 months. The patients already in the TolaSure Gel, 5% w/w cohort will continue with daily IP application for an additional 2 months as well. Again, patients have the option to continue to treat their feet. At Part 2 End of Study (EOS), patients will cease IP application and EOS procedures will be completed. Patients can have optional perilesional biopsies taken from a treated and untreated area to evaluate changes in ultrastructural pathology. A patient follow-up visit will occur after 6 months (2-months after last treatment application).

The primary endpoint will assess changes in disease severity within the TLAs and recurrence of blistering using clinical imaging to assess blister surface area over time. The secondary efficacy endpoints will evaluate blistering on the feet, subject self-assessments including pain, itch, modified Foot Function Index (mFFI), and Quality of Life (QoL) assessment.

Safety endpoints will include the incidence of treatment-emergent adverse events (TEAEs). In order to provide adequate assurance of subject safety, safety monitoring will include physical exams, vital sign measurements, clinical laboratory testing (blood and urinalysis), and urine pregnancy testing (as appropriate). These safety assessments in addition to adverse event (AE) reviews will be sufficient to identify potential TEAEs.

The information obtained from these assessments will be utilized to examine the efficacy of TolaSure treatment in ameliorating EBS symptoms as well as the accuracy of the proposed mechanism of action (MOA) of TolaSure for this disease indication.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or female at least 4 years of age.
* Patient has a documented diagnosis of generalize intermediate (previously Kӧbner) to severe (previously EBS-DM) autosomal dominant epidermolysis bullosa simplex (EBS) and/or genetic mutation in either the K14 or K5 genes consistent with generalized intermediate to severe EBS. The Investigator will determine patient eligibility based on historical phenotypic presentation of EBS symptoms along with genetic/diagnosis documentation in order to determine EBS severity. (If generalized intermediate to severe EBS is suspected but not diagnosed or genetically confirmed, confirmatory testing will be performed).
* Patient is actively flaring in one of the preferred target lesional areas (TLAs): 1) lower extremities (ideally below the knee and above the ankle or between the knee and top of the thigh) or 2) torso (excluding the groin and apocrine areas). The following skin conditions are required for treatment purposes:

  * A flare is defined as a minimum area of ~2-3% Body Surface Area (BSA) containing intact blisters (of varying size and number), and freshly ruptured blisters across 50% of the TLA (as assessed by the principal investigator (PI)). Skin erosions, keratoderma, fissures and/or erythema may also be present.
  * Patients will be permitted to treat their feet to assess plantar blister surface area but blistering on the feet is not a requirement for study inclusion.
  * TLA may not be infected (as assessed by PI) or have been treated with a topical antibiotic within 14 days.
* If the patient is a woman of childbearing potential (WOCBP),

  * Has a negative urine pregnancy test.
  * Agrees to use an approved effective form of birth control with failure rates <1% per year (e.g., implant, injectable, combined oral contraceptive, intrauterine contraceptive device, sexual abstinence, vasectomized partner) during participation in the study (and at least 3 months thereafter).
  * Is not nursing.
* Patient's laboratory values (blood and urine) are within the range of normal or abnormal values are within normal levels for the disease and in the opinion of the PI the values are not clinically relevant for study participation.
* Patient is in good, general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of the EBS lesions or which exposes the subject to an unacceptable risk by study participation.
* Over the duration of the study, the patient agrees to not use any other topical therapies and/or impregnated dressings within the TLAs (e.g., medicated cleansers, CBD oil, MediHoney, Silvadine cream 1%, topicals containing antimicrobials, keratin, and/or collagen, lipido-colloid or polymeric membrane dressings, and/or hydrogels).
* Patient and/or legally appointed and authorized representative must be able and willing to follow study procedures and instructions in order to maintain compliance throughout the study period.
* The patient or legally appointed and authorized representative must have read, understood and signed an Institutional Review Board/Ethics Committee (IRB/EC) approved Informed Consent or Assent Form.

Exclusion Criteria:

* Patient's use of prior or concomitant medication or medical treatments/procedures:

  * Any investigational drug or therapy within 30 days.
  * Systemic steroidal therapy within 30 days.
  * Topical steroidal therapy within 14 days (Note: inhaled and ophthalmic products containing steroids are allowed).
  * Systemic antibiotic therapy within 7 days.
  * Currently receiving chemotherapy or radiation.
  * Surgery within the previous 2 weeks (except for minor surgery, cosmetic or dental procedures as determined by the investigator).
  * Started to take chronic medications (NSAIDs, antihistamines, etc.) at least 30 days prior to starting study medication.
* Patient's medical history includes:

  * Cancer that is currently undergoing treatment.
  * History of chronic and severe vitamin, mineral, or protein deficiency.
  * Current systemic infection.
  * HIV/AIDS.
  * Non-EBS skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or condition (e.g., sunburn) that, in the opinion of the investigator, might put the patient at undue risk by study participation or interferes with the study medication application or the study assessments.
  * An illness (e.g., neurological, cardiovascular, respiratory, hepatic, renal, or metabolic disease), condition, or situation that in the opinion of the principal investigator is likely to interfere with the patient's participation in or completion of the study.
* Factors present in the patient and/or his/her legal representative that could interfere with study compliance such as inability to attend scheduled study visits or to perform study protocol procedures.
* Patient is a member of the investigational team or his/her immediate family.
* Other unspecified reasons that, in the opinion of the Investigator, make the patient unsuitable for enrollment.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Blister Surface Area of the Designated Treatment Area(s) | Day 1 (Baseline) and weekly until End of Study (2-months and maximum 4-months)
  Clinical photography will be used to assess changes in disease severity within the target lesional area (TLA) and recurrence of blistering by measuring blister surface area in the designated TLA over time.

SECONDARY OUTCOMES:
Plantar Blister Surface Area Reduction | Day 1 (Baseline) and weekly until End of Study (2-months and maximum 4-months)
  Plantar blister surface area changes over time will be examined using clinical photography for those patients that choose treat their feet. This is an optional treatment area.
Subject-reported Pain Score in Target Lesional Areas During Treatment Application | Day 1 (Baseline) and weekly until End of Study (2-months and maximum 4-months)
  Using the adult or pediatric PROMIS® Measure form, peak pain during treatment application will be reported on a weekly basis until Part 2 End of Study (EOS, 4-months), with a possible assessment at the 6-month follow up visit. Pain trends in TolaSure Gel, 5% w/w and Placebo groups will be compared. The following PROMIS® Measure forms will be used depending on the patient's age: The Adult Pain Interference-Short Form 8a, Pediatric Pain Interference-Short Form 8a, and Parent Proxy Pain Interference-Short Form 8a. These scales are from 1 to 5 and relate to how much pain interferes with daily activities, with 1 indicating Never/Not at All and 5 indicating Almost Always/Very Much.
Subject-reported Itch Score in Target Lesional Area | Day 1 (Baseline) and weekly until End of Study (2-months and maximum 4-months)
  Using the adult or pediatric PROMIS® Measure form, itch characteristics will be reported on a weekly basis until Part 2 End of Study (EOS, 4-months), with a possible assessment at the 6-month follow up visit. Itch trends in TolaSure Gel, 5% w/w and Placebo groups will be compared. The following PROMIS® Measure forms will be used depending on the patient's age: The Adult Itch Interference-Short Form 8a, Pediatric Itch-Short Form 8a (PIQ-C), and Parent Proxy Itch-Short Form 8a (PIQ-C). These scales are from 1 to 5 and relate to how much itch interferes with daily activities and the level of itch, with 1 indicating Never/No Itch and 5 indicating Almost Always/Very Severe.
Subject-reported Quality of Life (QoL) | Day 1 (Baseline), Part 1 End of Study (2-months), Part 2 End of Study (4-months)
  Patient's quality of life (QoL) metrics, highlighting symptoms and daily living concerns of EBS patients, will be reported at Visit 2/ Baseline, Part 1 End of Study (EOS), and Part 2 EOS, with a possible assessment at the 6-month follow up visit. This QoL assessment will be given to patients in a questionnaire format. The questions focus on how EBS blistering areas affect daily physical and social activities as well as mental and emotional health. The scale range is from 0 to 10, with 0 being not at all affected and 10 being severely affected. QoL metrics in TolaSure Gel, 5% w/w and Placebo control groups will be examined.
Subject-reported Modified Foot Function Index (mFFI) | Day 1 (Baseline), Part 1 End of Study (2-months), Part 2 End of Study (4-months)
  Patient's modified Foot Function Index (mFFI), is a questionnaire about foot pathology as it relates to pain, disability, and/or activity restrictions. Questions relating to pain are on a 0 to 10 scale with 0 being no pain at all and 10 being the worst pain imaginable. Daily activity scores also range from 0 to 10 with 0 being Not at All/Not Difficult at All and 10 being All the Time/So Difficult. The mFFI questionnaire will be reported at Visit 2/ Baseline, Part 1 End of Study (EOS), and Part 2 EOS, with a possible assessment at the 6-month follow up visit. mFFI metrics in TolaSure Gel, 5% w/w and Placebo control groups will be examined.
Incidence of treatment-emergent adverse events (TEAEs) | Day 1 (Baseline) and bi-weekly until End of Study (maximum 4-months)
  Safety monitoring will include clinical laboratory testing (blood and urine) and urine pregnancy testing (as appropriate) only at Visit 1/Screening and Part 2 EOS, physical examinations (including assessment of treatment areas), and vital sign measurements at baseline and bi-weekly until Part 1 EOS and Part 2 EOS. These assessments along with AE reviews will identify potential TEAEs.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Dermatology Department, Palo Alto, California
  - NU Dermatolgy CTU, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BioMendics, LLC — https://www.biomendics.com
- See also: Stanford Medicine, Dermatology, Current EB Studies — https://med.stanford.edu/dermatology/research/research_1/currentstudies.html
- See also: Northwestern Medicine, Department of Dermatology Clinical Trials — https://www.feinberg.northwestern.edu/sites/dermatology/research/clinical-trials.html